CLINICAL TRIAL: NCT03190096
Title: Safety and Feasibility of Electrical Isolation of the Superior Vena Cava in Addition to Pulmonary Vein Ablation for Paroxysmal Atrial Fibrillation Using the Cryoballoon: the SAFE-SVC Study.
Brief Title: Safety and Feasibility of Electrical Isolation of the Superior Vena Cava for Paroxysmal Atrial Fibrillation
Acronym: SAFE-SVC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ettore Sansavini Health Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ESREFO 31
Record Dates: First submitted 2017-06-08; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: SVC isolation — After PVI ablation SVC will be performed. The CB will be retrieved to the right atrium and the achieve catheter will be advanced in the SVC. The CB will be inflated in the right atrium and advanced towards the ostium of the SVC to occlude the vessel

SUMMARY:
The present study is designed as a observational prospective, multicentre, international. The main aim of this study is to evaluate the safety and feasibility of SVC isolation with the CB in a prospective manner.

DETAILED DESCRIPTION:
Consecutive patients programmed for cryoballoon ablation (CBA) for PAF will be prospectively enrolled in our study. After PVI is obtained and proven by entrance- and exit block, the SVC will be mapped for potentials. If the SVC exhibits electrical activity, isolation will be attempted performing a single maximum 180 seconds balloon application. A single 180 seconds application is known to produce a durable lesion. Performing a combined approach (PVI together with SVC isolation) using the same cryoballoon requires no additional vascular access. Therefore no significant raise in complications is to be expected. During a second generation CBA the described rate of complications is to be estimated around 2%. Transient phrenic nerve palsy in 7.2 %, but reversible in virtually all patients within the end of the procedure.

To prevent nervous injury the phrenic nerve (PN) will be tested during ablation of the SVC, in the same fashion as performed systematically during ablation of the right sided pulmonary veins.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Consecutive patients programmed for cryoballoon ablation (CBA) for PAF will be prospectively enrolled in our study

Exclusion Criteria:

1. Age younger than 18 years
2. Severe valve disease (MI or AI > ¾)
3. Uncontrolled heart failure,
4. Contraindication to general anaesthesia/ deep procedural sedation
5. Left atrial thrombus at the pre-procedural transesophageal echocardiogram (TEE)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients programmed for cryoballoon ablation (CBA) for PAF
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-06-07 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
SVC isolation using a dedicated cryoballoon device | During procedure
  feasibility and safety of superior vena cava (SVC) isolation added to standard pulmonary vein isolation using the cryoballoon in patients with paroxysmal atrial fibrillation

SECONDARY OUTCOMES:
Clinical outcame | 12 months
  Clinical outcome in terms of freedom from atrial fibrillation following ablation.

OTHER OUTCOMES:
Clinically relevant abnormalities | 12 months
  Detection of clinically relevant abnormalities on physical examinations, vital signs, 2D echocardio, 12 lead ECG, and laboratory routine tests.

CONTACTS AND LOCATIONS:
Overall Officials: Saverio Iacopino, MD, Principal Investigator — Maria Cecilia Hospital
Locations (4):
- UZ Brussel VUB, Brussels, Belgium
- Maria Cecilia Hospital, Cotignola, Ravenna, Italy
- Radboud University, Nijmegen, Netherlands
- Novosibirsk University, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No